CLINICAL TRIAL: NCT05673850
Title: Association Between HER2 Status and pCR Rate in ER-positive Breast Cancer Receiving Neoadjuvant Endocrine or Chemotherapy
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: ASSOCIHER
Record Dates: First submitted 2022-11-27; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-11

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NET
  Interventions: Drug: NET or NCT
- NCT
  Interventions: Drug: NET or NCT

INTERVENTIONS:
Drug: NET or NCT — In this study, we included 518 ER-positive BC patients who received either neoadjuvant endo-crine therapy (NET) or neoadjuvant chemotherapy (NCT).

SUMMARY:
In estrogen receptor (ER)-positive breast cancer (BC), human epidermal growth factor receptor-2 (HER2)-low ones are reported to have distinct clinical and molecular features from those with HER2-zero or HER2-positive status. However, the association between HER2-low status with response to endocrine therapy is largely unknown. In this study, we included 518 ER-positive BC patients who received either neoadjuvant endocrine therapy (NET) or neoadjuvant chemotherapy (NCT). The pathologic complete response rate (pCR) of HER2-low and HER2-zero tumors re-sponding to neoadjuvant therapies were compared. The difference in disease-free survival (DFS) and overall survival (OS) between the two groups was also analyzed. The pCR (defined as ypT0/isNx) in HER2-low BCs and in HER2-zero BCs for NET cohort and NCT cohort were compared.

ELIGIBILITY:
Inclusion Criteria:

patients diagnosed with invasive breast cancer and who received surgery from 2015 to 2021

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In this retrospective cohort study, we sourced data from the electronic database of Peking university cancer hospital to identify patients diagnosed with invasive breast cancer and who received surgery from 2015 to 2021. Patients were excluded by the fol-lowing criteria: (1) patients who were ER-negative; (2) patients who were HER2 posi-tive defined as IHC3+ or IHC2+/fluorescence in situ hybridization (FISH)-positive; (3) patients who were HER2 (IHC2+) but did not evaluate by further FISH;(4) patients who did not receive neoadjuvant therapy; (5) patients who received concurrent neo-adjuvant endocrine and chemotherapy. Patients who remained were further divided into two groups: those receiving neoadjuvant endocrine therapy (the NET group) and those receiving neoadjuvant chemotherapy (the NCT group).
Sampling Method: Non-Probability Sample
Enrollment: 518 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
pathologic complete response rate (pCR) | through study completion, an average of 6 months
  ypT0/isNx

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Haidian, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No